CLINICAL TRIAL: NCT02428088
Title: A 6-week, Randomized, Double-Blind, Multicenter, Placebo-Controlled, Parallel-group Efficacy and Safety Study of Dasotraline Versus Placebo in Subjects 6 to 12 Years of Age With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Dasotraline Pediatric ADHD Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEP360-202
Record Dates: First submitted 2015-04-20; First posted 2015-04-28 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 4-(3,4-dichlorophenyl)-1,2,3,4-tetrahydronaphthalen-1-amine; SEP 225289

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dasotraline 2 mg (Experimental): Dasotraline 2 mg
  Interventions: Drug: Dasotraline
- Dasotraline 4 mg (Experimental): Dasotraline 4 mg
  Interventions: Drug: Dasotraline
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Dasotraline — Dasotraline 2 mg once daily
  Other Names: SEP-225289
  Arms: Dasotraline 2 mg
Drug: Dasotraline — Dasotraline 4 mg once daily
  Other Names: SEP-225289
  Arms: Dasotraline 4 mg
Drug: Placebo Comparator — Placebo once daily
  Arms: Placebo

SUMMARY:
This is a 6 week efficacy and safety study of Dasotraline in subjects 6 to 12 years old with ADHD.

DETAILED DESCRIPTION:
This is a randomized, double blind, multicenter, placebo-controlled, parallel group, outpatient study evaluating the efficacy and safety of dasotraline in subjects 6 to 12 years of age with ADHD using 2 doses of dasotraline (2 mg/day and 4 mg/day) versus placebo over a 6 week treatment period. The study will consist of screening, treatment, and end of study visits.

ELIGIBILITY:
Inclusion Criteria:

* Subject's parent/legal guardian must give written informed consent, including privacy authorization, prior to study participation. The subject will complete an informed assent prior to study participation.
* Subject and the subject's parent/legal guardian must be judged by the investigator to be willing and able to comply with the study procedures and visit schedules.
* Subject, male or female, must be between 6 and 12 years of age, inclusive, at the time of consent/assent and at Baseline.
* Subject meets Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM 5) criteria for a primary diagnosis of ADHD (inattentive, hyperactive, or combined presentation) at screening established by a comprehensive psychiatric evaluation that reviews DSM 5 criteria is confirmed using the K-SADS-PL at Screening.
* Subject has an ADHD RS IV HV score of ≥ 28.
* Subject has a CGI S score of ≥ 4.
* Subject, if female, must not be pregnant or breastfeeding, and if ≥ 8 years of age must have a negative pregnancy test.
* Female subject:

  * must be unable to become pregnant (eg, premenarchal, surgically sterile, etc);

OR

• practice true abstinence (consistent with lifestyle) and must agree to remain abstinent from signing informed consent/assent to at least 14 days after the last dose of study drug has been taken;

OR

• is sexually active and willing to use a medically effective method of birth control (see Appendix VII) from signing informed consent/assent to at least 14 days after the last dose of study drug has been taken.

* Male subject must be willing to remain sexually abstinent (consistent with lifestyle) or be using an effective method of birth control from signing informed consent/assent to at least 14 days after the last dose of study drug has been taken.
* Subject must be in general good health (defined as the absence of any clinically relevant abnormalities as determined by the Investigator) based on screening physical and neurological examinations, vital signs, medical history, and clinical laboratory values (hematology, chemistry, and urinalysis). Note: If any of the hematology, chemistry, or urinalysis results are not within the laboratory's reference range, then the subject may be included only if the investigator determines the deviations to be not clinically relevant.
* Subject weighs at least 21 kg and is within 3rd to 97th percentile for gender specific body-mass-index (BMI)-for-age from the World Health Organization (WHO) growth charts (see Appendices II and IX).
* Subject's parent/legal guardian must report a history of the subject being able to swallow capsules.
* Subject and subject's parents/legal guardians must be able to fully comprehend the informed consent/assent form (as applicable), understand all study procedures, and be able to communicate satisfactorily with the Investigator and study coordinator.

Exclusion Criteria:

* Subject or parent/legal guardian has commitments during the study that would interfere with attending study visits.
* Subject currently has a diagnosis of asthma that has required daily treatment with bronchodilators or nebulizer treatments in the 30 days prior to screening and/or who may require daily treatments with these agents over the course of the trial. Intermittent use of bronchodilators is not exclusionary. Subjects who have a history of requiring persistent asthma treatment should be discussed wit the medical monitor prior to enrolment.
* Subject has any clinically significant unstable medical abnormality, chronic disease, or a history of a clinically significant abnormality of the cardiovascular, gastrointestinal, respiratory, hepatic, or renal systems, or a disorder or history of a condition (eg, malabsorption, gastrointestinal surgery) that may interfere with drug absorption, distribution, metabolism, or excretion. Note: Active medical conditions that are minor or well-controlled are not exclusionary if they do not affect risk to the subject or the study results. In cases in which the impact of the condition upon risk to the subject or study results is unclear, the Medical Monitor should be consulted. Any subject with a known cardiovascular disease or condition (even if controlled) must be discussed with the Medical Monitor during screening.
* Subject has a history or presence of abnormal ECGs, which in the investigator's opinion is clinically significant. Screening site ECGs will be centrally over-read, and eligibility will be determined by the investigator based on the results of the over-read report.
* Subject has any documented diagnosis of Bipolar I or II Disorder, major depressive disorder, conduct disorder, obsessive-compulsive disorder, disruptive mood dysregulation disorder (DMDD), intellectual disability, any history of psychosis, autism spectrum disorder, Tourette's Syndrome, confirmed genetic disorder with cognitive and/or behavioral disturbances. Note: Subjects with oppositional defiant disorder (ODD) are permitted to enroll in the study as long as ODD is not the primary focus of treatment.
* Subject has generalized anxiety disorder that has been the primary focus of treatment at any time during the 12 months prior to screening or that required pharmacotherapy any time in the 6 months prior to screening.
* Subject has failed 2 adequate courses of stimulant or non-stimulant treatment for ADHD, as judged by the investigator.
* Subject has evidence of any chronic disease of the central nervous system (CNS) such as tumors, inflammation, seizure disorder, vascular disorder, potential CNS related disorders that might occur in childhood (eg, Duchenne Muscular dystrophy, myasthenia gravis, or other neurologic or serious neuromuscular disorders), or history of persistent neurological symptoms attributable to serious head injury. Past history of febrile seizure, drug-induced seizure, or alcohol withdrawal seizure is exclusionary. Subject taking anticonvulsants for seizure control currently or within the past 2 years is not eligible for study participation.
* Subject has uncontrolled thyroid disorder indicated by free T4, free T3, or thyroid stimulating hormone (TSH) outside the limit of normal for the reference laboratory.
* Subject answers "yes" to "Suicidal Ideation" item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) for any lifetime history on the C SSRS Children's Lifetime/Recent assessment at screening.
* Subject has any history of attempted suicide, in the opinion of the investigator.
* Subject does not tolerate venipuncture or has poor venous access that would cause difficulty for collecting blood samples.
* Subject has a history of severe allergies to more than 1 class of medications or multiple adverse drug reactions or has a history of allergic reaction or has a known or suspected sensitivity to any substance that is contained in the study drug formulations.
* Subject has history of intolerance to stimulants.
* Subject has taken any antipsychotic medication within 8 weeks prior to screening.
* Subject taking any medication, including health food supplements with purported psychotropic activity (for example, St. John's Wort), must have a minimum washout of 7 days prior to Day 1.
* Subject taking any antidepressant medication (eg, bupropion, selective serotonin reuptake inhibitor [SSRI]/ serotonin norepinephrine reuptake inhibitor [SNRI], monoamine oxidase [MAO] inhibitor, tricyclic, etc) must have a minimum washout of 7 days prior to Day 1.
* Subject is currently undergoing Cognitive Behavioral Therapy (CBT) for the treatment of ADHD, has initiated behavioral therapy (including school based interventions) less than 1 month prior to screening, or is receiving behavioral therapy and in the opinion of the investigator will not be able to follow a stable routine for the duration of the study.
* Subject or subject's family anticipates a move outside the geographic range of investigative site during the study period, or plans extended travel inconsistent with the recommended visit interval during study duration.
* Subject has a history of, or current malignancy except for non melanomatous skin cancer.
* Subject has history of positive test for Hepatitis B surface antigen or Hepatitis C antibody and has liver function test results at screening above the upper limit of normal for the reference laboratory.
* Subject is known to have tested positive for human immunodeficiency virus (HIV).
* Subject has participated in any investigational study within 90 days prior to screening or is currently participating in another clinical trial.
* Subject has a history of substance or alcohol use disorder (excluding caffeine) within the 12 months prior to screening, as defined by the DSM 5 criteria, or is currently using tobacco or other nicotine-containing products, or has a positive urine drug screen (UDS) or breath alcohol test at screening. Note: Subjects with a positive UDS may be allowed to continue in the study, provided that the investigator determines that the positive test is as a result of taking prescription medicine(s) as prescribed.
* Subject requires treatment with any disallowed medications during the study.
* Subject has experienced significant blood loss within 60 days prior to screening.
* Subject has previously been enrolled in a clinical trial of dasotraline (SEP 225289).
* Subject's parent/legal guardian is an investigational site staff member or the relative of an investigational site staff member.
* Subject is, in the opinion of the Investigator, unsuitable in any other way to participate in this study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 330 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline at Week 6 in ADHD symptoms as measured by ADHD RS IV HV. | Baseline, 6 Weeks

SECONDARY OUTCOMES:
Change from baseline in ADHD symptoms as measured by in ADHD RS IV HV at Weeks 1, 2, 3, 4, and 5. | Baseline, Weeks 1,2,3,4,5
Change from baseline in the inattentiveness and hyperactivity subscales of the ADHD RS IV HV at Weeks 1, 2, 3, 4, 5, and 6. | Baseline, Weeks 1,2,3,4,5,6
The percentage of responders at Weeks 1, 2, 3, 4, 5, and 6. A responder is defined as a subject with a ≥ 30% improvement in ADHD symptoms compared with baseline as measured by the ADHD RS IV HV. | Baseline, Weeks 1,2,3,4,5,6
Change from baseline in CGI-S scale at Weeks 1, 2, 3, 4, 5, and 6. | Baseline, Weeks 1,2,3,4,5,6
Change from baseline in Conners 3 P total score and subscale scores (Oppositional, Cognitive problems, Hyperactivity, and ADHD Index) at Weeks 1, 2, 3, 4, 5, and 6. | Baseline, Weeks 1,2,3,4,5,6
Change from baseline in Conners 3 T total score at Weeks 3 and 6. | Baseline, Weeks 3, 6
Change from baseline in WPREMB R total score and subscores at Weeks 1, 2, 3, 4, 5, and 6. | Baseline, Weeks 1,2,3,4,5,6
The incidence of overall AEs, serious AEs (SAEs), and AEs (or SAEs) leading to discontinuations. | Baseline, 6 Weeks
Absolute values and change from baseline in clinical laboratory evaluations (serum chemistry). | Baseline, 6 Weeks
Absolute values and change from baseline in clinical laboratory evaluations (hematology). | Baseline, 6 Weeks
Absolute values and change from baseline in clinical laboratory evaluations (lipid panel). | Baseline, 6 Weeks
Absolute values and change from baseline in clinical laboratory evaluations (thyroid panel). | Baseline, 6 Weeks
Absolute values and change from baseline in clinical laboratory evaluations (sex hormones). | Baseline, 6 Weeks
Absolute values and change from baseline in clinical laboratory evaluations (urinalysis). | Baseline, 6 Weeks
Absolute values and changes from baseline in 12 lead ECGs. | Baseline, 6 Weeks
Absolute values and changes from baseline in vital signs. | Baseline, 6 Weeks
Absolute values and changes from baseline in body weights. | Baseline, 6 Weeks
Change from baseline in CSHQ total score and 8 subscale scores (bedtime resistance, sleep onset delay, sleep duration, sleep anxiety, night wakings, parasomnias, sleep disordered breathing, and daytime sleepiness) at Weeks 1, 2, 3, 4, 5, and 6. | Baseline, Weeks 1,2,3,4,5,6
Change from baseline in Tanner staging at Week 6. | 6 Weeks
Frequency of suicidal ideation and suicidal behavior as assessed by the C SSRS. | 6 Weeks
Severity of suicidal ideation and suicidal behavior as assessed by the C SSRS. | 6 Weeks
Dasotraline plasma concentration for PK at Weeks 2, 4, and 6. | Baseline, Weeks 2,4,6
Change from baseline in DHPG concentration at Weeks 2, 4, and 6. | Baseline, Weeks 2,4,6
Change from baseline in NE concentration at Weeks 2, 4, and 6. | Baseline, Weeks 2,4,6
Change from baseline in WFIRS P total score and 6 domain scores (family, learning and school, life skills, child's self-concept, social activities and risky activities) at Week 3 and 6. | Baseline, Weeks 3,6

CONTACTS AND LOCATIONS:
Overall Officials: Dasotraline Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (43):
- United States (43):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Synergy Research, National City, California
  - California Clinical Trials, Paramount, California
  - PCSD-Feighner Research, San Diego, California
  - Elite Clinical Trials, Inc., Wildomar, California
  - MCB Clinical Research Centers, LLC, Colorado Springs, Colorado
  - Gulfcoast Clinical Research, Fort Myers, Florida
  - Sarkis Clinical Trials - Parent, Gainesville, Florida
  - Palm Springs Research Institute, Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Capstone Clinical Research, Inc., Libertyville, Illinois
  - Baber Research Group, Naperville, Illinois
  - Goldpoint Clinical Research, Indianapolis, Indiana
  - Pedia Research,LLC, Newburgh, Indiana
  - Psychiatric Associates, Overland Park, Kansas
  - Pedia Research,LLC, Owensboro, Kentucky
  - Hugo W. Moser Research Institute at Kennedy Krieger, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Neurobehaviorial Medicine Group, PLLC, Bloomfield Hills, Michigan
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - Midwest Research Group, Saint Charles, Missouri
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Pharmaceutical Research Associates, Inc., Marlton, New Jersey
  - Richmond Behavioral Associates, Staten Island, New York
  - Duke University Medical Center - Duke Child and Family Study Center, Durham, North Carolina
  - University of Cincinnati/Department of Psychiatry and Behavioral Neuroscience, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - North Star Medical Research, LLC, Middleburg Heights, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Cyn3rgy Research, Gresham, Oregon
  - BioBehavioral Research of Austin P.C., Austin, Texas
  - Pillar Clinical Research, LLC, Dallas, Texas
  - Bayou City Research Corporation, Houston, Texas
  - Houston Clinical Trials, LLC, Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Road Runner Research, San Antonio, Texas
  - Family Psychiatry of The Woodlands, P.A., The Woodlands, Texas
  - Aspen Clinical Research, Orem, Utah

REFERENCES:
- [Derived] Findling RL, Adler LA, Spencer TJ, Goldman R, Hopkins SC, Koblan KS, Kent J, Hsu J, Loebel A. Dasotraline in Children with Attention-Deficit/Hyperactivity Disorder: A Six-Week, Placebo-Controlled, Fixed-Dose Trial. J Child Adolesc Psychopharmacol. 2019 Mar;29(2):80-89. doi: 10.1089/cap.2018.0083. Epub 2019 Jan 29. PMID 30694697